CLINICAL TRIAL: NCT04714957
Title: PITCHER (Peritoneal Carcinomatosis Heterogeneity)
Status: Recruiting | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL16_0672
Record Dates: First submitted 2021-01-14; First posted 2021-01-20 (Actual); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Secondary Peritoneal Cancers; Colorectal Cancer; Ovarian Cancer
Keywords: peritoneal carcinomatosis; tumor heterogeneity; epigenetic landscape
MeSH Terms: conditions — Colorectal Neoplasms; Ovarian Neoplasms; Peritoneal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor samples (peritoneal carcinomatosis, primary tumor, other tumor metastasis (when applicable)), healthy tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: construction of a database of genetic and epigenetic data on peritoneal carcinomatosis of colorectal or ovarian origin. — Construction of a core database of genetic and epigenetic markers, in order to identify predictive biomarkers and potentially actionable targets for controlling the spread of peritoneal carcinomatosis.

SUMMARY:
How epigenetic deregulation affects gene expression patterns in subclones of the same tumor is poorly known. Peritoneal Carcinomatosis (PC) is a condition in which multiple metastases of the same abdominal tumor develop in the peritoneal cavity and intra-peritoneal organs, thus defining different ecosystems of the same cancer. PITCHER addresses the variations in epigenetically regulated gene expression between different subclones of PC in relation with cell mechanoresponses, providing insights on how cancer epigenetic landscapes evolve under environmental pressures and on strategies used by cancer cells to adapt to the transition from one ecosystem to the other.

PITCHER is a network of 10 teams from Lyon, Grenoble and Marseille, based on data and specimen collection of patients who have undergone a surgery for a peritoneal carcinomatosis of ovarian or colorectal origin. PC lesions and eventually matched specimens of primary tumors will be collected in the same patients at the time of the surgery or eventually retrieved from already existing samples. Epigenetic landscapes will be analyzed by a bioinformatics pipeline combining exome sequencing, transcriptome and methylome to identify "epigenetic hotspots", and their variations across lesions will be evaluated. These analyses will be realized in fresh (when available) or pre-existing samples. When possible, organoid cultures and animal models will be derived from multicellular structures in peritoneal fluids and membrane, cytoskeletal and nucleoskeletal mechanoresponses will be characterized using Atomic Force Microscopy. The role of tumor axonogenesis, a process of neo-formation of axon fibers in tumors, will be addressed. Experimental studies of cell responses to therapy will be performed to derive mathematical predictive models. All components will be integrated in a systems biology map of PC.

ELIGIBILITY:
Inclusion Criteria:

* Patients who accept to participate to the study
* Men / women aged over 18 years
* Patients with cancer management and care for peritoneal carcinomatosis of digestive or ovarian origin
* Patients had histologic/radiologic confirmation of peritoneal disease
* Serology negative HIV, HEPATITIS

Exclusion Criteria:

• none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cancer management and care for peritoneal carcinomatosis of digestive or ovarian origin. PITCHER will include patients who will undergo surgery for peritoneal carcinomatosis or patients who already undergone surgery for peritoneal carcinomatosis
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
genetic and epigenetic data available for 20 "multiplets" biospecimens (peritoneal carcinomatosis + healthy tissue + primary tumor + tissue from other tumor metastasis - when applicable and available- ) | end of the inclusion period (September 2022)
  The main endpoint is to implement a specific tissue collection of appropriate quality, assembling "multiplets" of biospecimens from the same patient, in order to construct a core database for research on mechanisms, biomarkers and actionable therapeutic targets in PC. This database will include molecular analysis by next-generation sequencing of whole-exome genetic, transcriptomic and epigenetic patterns of primary, peritoneal and metastatic lesions. "Omics" data are compiled using a data model also including anonymized information on histopathology and clinical history of treatments (when applicable)

CONTACTS AND LOCATIONS:
Locations (1):
- Lyon SUD Hospital, Hospices Civils de Lyon, Lyon, France